CLINICAL TRIAL: NCT05853393
Title: Sleep and Eating Behaviors in Rural Preadolescent Children (Tween SPACE [Sleep Patterns, Appetite Control, and Environment])
Brief Title: Tween Sleep Patterns, Appetite Control, and Environment
Acronym: TweenSPACE
Status: Completed | Type: Observational
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Emily Hohman, Assistant Research Professor, Penn State University
Other Study IDs: STUDY00020663
Record Dates: First submitted 2023-04-21; First posted 2023-05-10 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Child Obesity; Eating Behavior; Sleep
Keywords: sleep; eating in the absence of hunger; eating; preadolescent; rural; actigraphy; ecological momentary assessment
MeSH Terms: conditions — Pediatric Obesity; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this study is to learn about how children's sleep is related to their eating behaviors the next day, and to learn about factors that relate to eating behaviors and sleep health that are specific to preadolescent children living in rural communities.

DETAILED DESCRIPTION:
The aims of this study are to a) describe the prevalence and characteristics of eating in the absence of hunger (EAH) in rural preadolescent children using a novel methodology, ecological momentary assessment (EMA); b) to examine the within-person temporal relationship between daily changes in sleep health (i.e., duration and quality) and EAH; and c) examine associations between family, child, and environmental characteristics, sleep, and eating behaviors in rural preadolescent children. Parent-child dyads will participate in the study via remote data collection methods including Zoom interviews, online surveys, EMA survey completed by smartphone, and actigraphy.

ELIGIBILITY:
Child Inclusion Criteria:

1. Age 8 to 12 years
2. Primary residence is in a rural ZIP code in the United States, as defined by Health Resources & Services Administration
3. BMI for age ≥ 85th percentile OR BMI ≥ 15th percentile plus at least one biological parent with BMI ≥ 25 kg/m2
4. Able to read and answer questions in English

Parent Inclusion criteria:

1. Parent or caregiver of an eligible child
2. Age 18 years or older
3. Able to read and answer questions in English

Exclusion Criteria:

1. Any medical condition that significantly impacts eating, sleep, growth, or ability to operate the mEMA smartphone platform (e.g., eating disorder, Type I diabetes, blindness) (Child participants only)
2. Unable to connect to a Zoom session via internet or cell-phone data from home
3. Unable to receive and sign for package with study supplies

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children 8-12 years old and a parent/guardian (n=64 parent-child dyads for a total of 128 individuals)
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of eating in the absence of hunger (EAH) episodes | Multiple measurements per day for 2 weeks starting at enrollment through 2 weeks
  Eating events where pre-meal hunger is less than 35 on a 100 point visual analogue scale, as reported on smartphone surveys that are completed multiple times a day over a 2 week period.

SECONDARY OUTCOMES:
Visual analogue scale rating of hunger | Multiple measurements per day for 2 weeks
  Collected via EMA
Visual analogue scale rating of fullness | Multiple measurements per day for 2 weeks
  Collected via EMA
Visual analogue scale rating of desire to eat | Multiple measurements per day for 2 weeks
  Collected via EMA
Child appetitive traits | At enrollment
  Measured by parent report questionnaire (Child Eating Behavior Questionnaire)
Child mindful eating | At enrollment
  Measured by child self report questionnaire (Mindful Eating Questionnaire)
Child eating motivations | At enrollment
  Measured by child self report questionnaire (Palatable Eating Motives Questionnaire)
Child restrained and disinhibited eating | At enrollment
  Measured by child self report questionnaire (Dutch Eating Behavior Questionnaire)
Sleep duration | Daily over 2 weeks
  Measured by actigraphy
Sleep maintenance efficiency | Daily over 2 weeks
  Measured by actigraphy
Body mass index z-score | At enrollment
  Calculated from measured height and weight

CONTACTS AND LOCATIONS:
Overall Officials: Emily E Hohman, PhD, Principal Investigator — Penn State University
Locations (1):
- Pennyslvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified participant data may be made available at the conclusion of the study by request to the PI